CLINICAL TRIAL: NCT00416858
Title: Randomized Study of Adjuvant Radiochemotherapy After Surgery Versus Radiochemotherapy Alone in Patients With Locally Advanced Esophageal Cancer
Brief Title: Radiation Therapy and Combination Chemotherapy With or Without Surgery in Treating Patients With Locally Advanced Esophageal Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000453783; FFCD-9102; EU-20539; ESSAI-FFCD-9102
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2007-04

CONDITIONS: Esophageal Cancer
Keywords: stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Fluorouracil; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain.

PURPOSE: This randomized phase III trial is studying radiation therapy together with combination chemotherapy to see how well they work with or without surgery in treating patients with locally advanced esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with locally advanced esophageal cancer treated with neoadjuvant radiotherapy and chemotherapy comprising fluorouracil and cisplatin followed by surgery or radiotherapy and chemotherapy.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to gender, histology (epidermoid vs glandular), response to induction therapy (complete vs partial), and tumor differentiation (little differentiated vs undifferentiated/good vs moderately differentiated).

* Induction therapy: All patients receive induction therapy comprising fluorouracil IV continuously over 24 hours on days 1-5 and cisplatin IV over 1 hour on days 1-5 or on day 2. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo radiotherapy twice daily on days 1-5 and 22-26 or once daily 5 days a week for 4½ weeks. Patients achieving complete or partial response are randomized to 1 of 2 treatment arms.
* Arm I: Patients undergo surgery. Patients may receive 1 course of adjuvant chemotherapy (as in induction therapy) and undergo additional radiotherapy.
* Arm II: Patients receive additional fluoroucacil and cisplatin as in induction therapy. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo additional radiotherapy once daily 5 days a week for 2 weeks.

Quality of life is assessed at baseline, after treatment on arms I or II, and then every 2 months (arm I) or every 6 months (arm II) thereafter.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed epidermoid or glandular cancer of the esophagus meeting the following criteria:

  * Tumor volume with or without mediastinal adenopathy, celiac, or subclavicular involvement
  * T3, N0-N1 disease
  * Tumor extends into fifth stratum by endosonographic scan
  * Resectable disease (palliative or curative)
* No cervical tumor
* No T1, T2, or T4 tumors
* No tracheo-esophageal fistula or tracheal invasion
* No gastric cardia cancer by gastroscopy
* No visceral (e.g., lung, bone, brain, liver), ganglion, or clavicular metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Creatinine normal
* WBC ≥ 3,000/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Transaminases ≥ 60%
* Bilirubin ≤ 2.0 mg/dL
* No cirrhosis
* DLCO ≥ 1.5 L with or without hypoxemia at rest
* No progressive coronary insufficiency
* Weight loss ≤ 15%
* No other malignancy in the past 2 years
* Must be able to maintain sufficient enteral nutrition (2,000 calories/day)

  * Laser photodestruction, dilation, or gastric balloon allowed
* No contraindication to radiotherapy
* No recurring left paralysis

PRIOR CONCURRENT THERAPY:

* No concurrent nephrotoxic or myelotoxic drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bedenne, MD, Study Chair — Federation Francophone de Cancerologie Digestive

REFERENCES:
- [Result] Burtin P, Bouche O, Giovannini M, Pelletier M, Conroy T, Ruget O, Arsene D, Milan C, Bedenne L. Endoscopic ultrasonography is an independent predictive factor of prognosis in locally advanced esophageal cancer. Results from the randomized FFCD 9102 study from the Federation Francophone de Cancerologie Digestive. Gastroenterol Clin Biol. 2008 Mar;32(3):213-20. doi: 10.1016/j.gcb.2007.12.026. Epub 2008 Mar 26. PMID 18372134
- [Result] Bedenne L, Michel P, Bouche O, Milan C, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Herr JP, Paillot B, Arveux P, Bonnetain F, Binquet C. Chemoradiation followed by surgery compared with chemoradiation alone in squamous cancer of the esophagus: FFCD 9102. J Clin Oncol. 2007 Apr 1;25(10):1160-8. doi: 10.1200/JCO.2005.04.7118. PMID 17401004
- [Result] Crehange G, Maingon P, Peignaux K, N'guyen TD, Mirabel X, Marchal C, Verrelle P, Roullet B, Bonnetain F, Bedenne L; Federation Francophone de Cancerologie Digestive 9102. Phase III trial of protracted compared with split-course chemoradiation for esophageal carcinoma: Federation Francophone de Cancerologie Digestive 9102. J Clin Oncol. 2007 Nov 1;25(31):4895-901. doi: 10.1200/JCO.2007.12.3471. PMID 17971585
- [Result] Bonnetain F, Bouche O, Michel P, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Paillot B, Arveux P, Milan C, Bedenne L. A comparative longitudinal quality of life study using the Spitzer quality of life index in a randomized multicenter phase III trial (FFCD 9102): chemoradiation followed by surgery compared with chemoradiation alone in locally advanced squamous resectable thoracic esophageal cancer. Ann Oncol. 2006 May;17(5):827-34. doi: 10.1093/annonc/mdl033. Epub 2006 Mar 8. PMID 16524973